CLINICAL TRIAL: NCT00631501
Title: Doxycycline for Lateral Epicondylalgia - RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaunas University of Medicine (Other)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Per Aspenberg, Dept of Orthopaedics, University Hospital Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BE-2-47
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2008-02

CONDITIONS: Lateral Epicondylalgia (Tennis Elbow)
Keywords: tendinopathy; tennis elbow; lateral epicondylitis; lateral epicondylalgia; MMP-inhibitor
MeSH Terms: conditions — Tennis Elbow; Tendinopathy | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Doxycycline (Experimental): 100 mg twice daily
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Placebo
  Arms: 2
Drug: Doxycycline
  Arms: Doxycycline

SUMMARY:
Matrix metalloproteinases are involved in the pathogenesis of tendinopathy. Doxycycline, a widely available pharmaceutical agent mostly used for its antibiotic properties, also functions as an inhibitor of MMPs.

This study aims to investigate the effect of doxycycline treatment on lateral epicondylalgia (tennis elbow). During three weeks, patients receive doxycycline tablets 100 mg twice daily, or placebo. Main outcome variable is pain (VAS) at three weeks.

Serum and/or plasma levels of matrix metalloproteinases and tissue inhibitors of metalloproteinases are measured.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Pain at the lateral side of the elbow ≥8 weeks
* Local tenderness on palpation of the lateral epicondyle
* Pain on resisted extension of the wrist

Exclusion Criteria:

* Rheumatic disorder
* History of fibromyalgia or generalised pain
* Elbow surgery (on the painful side)
* Active infection
* Glucocorticoid treatment during the duration of symtoms of epicondylalgia
* NSAID use within 1 w before presentation and during the study
* Pregnancy
* Taking drug that might interact with doxycycline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)

PRIMARY OUTCOMES:
Pain (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Orthopaedics, Kaunas Medical University, Kaunas, Kaunas County, Lithuania